CLINICAL TRIAL: NCT06556823
Title: Comparison of Contralateral Leg Neuro-dynamic Technique and Spine Mobilization With Leg Movement in Diabetic and Non-diabetic Patients With Sciatica
Brief Title: Contralateral Leg Neuro-dynamic and Spine Mobilization With Leg Movement in Patients With Sciatica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01864 Aiman Alam
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Sciatic Radiculopathy
Keywords: Contralateral leg neuro-dynamic technique,; Spine mobilization with leg movement; Sciatica due to lumbar degenerative problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Contralateral Leg Neuro Dynamic+ Conventional PT in Diabetic Population): (Experimental): The participant will be asked to sit on edge of table with hand behind the back with neutral spine. Then patient will be asked to adopted slump forward thoracic and lumbar spine. Then flex the patient neck passively and extend the patient asymptomatic knee with ankle dorsiflexion passively. Adopt this position for 30 sec and 12 rep will be perform for 3 sets and 4 rep per set.
  Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 10 min 2. Hot pack for 15 min 3. Bridging Exercises (10 rep x 1 Set with 3 sec hold) 4. Ankle pumps (10 rep x 1 Set).
  Interventions: Other: CLNDT+ Conventional PT in Diabetic Population):
- contralateral Leg Neuro Dynamic+ Conventional PT in non Diabetic Population): (Experimental): The patient will be asked to adopted slump forward thoracic and lumbar spine. Then flex the patient neck passively and extend the patient asymptomatic knee with ankle dorsiflexion passively. Adopt this position for 30 sec and 12 rep will be perform for 3 sets and 4 rep per set.
  Interventions: Other: CLNDT+ Conventional PT in non Diabetic Population):
- Spine Mobilization With Leg Movement+ Conventional PT in Diabetic Population) (Experimental): the participant will be asked to adopt side-lying position on their un-effected side, at edge of treatment table. Then The therapist will be applying transverse glide at spinous process towards floor. Other Therapist extended with slight abduction of 10 degrees and hip and knee flexed to 45 degrees. The participant will actively move into SLR with other therapist assistance. If participant feel pain, then ask them to breathe deeply and hold position for 3 sec.
  Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 10 min 2. Hot pack for 15 min 3. Bridging Exercises (10 rep x 1 Set with 3 sec hold) 4. Ankle pumps (10 rep x 1 Set)
  Interventions: Other: SMWLM+ Conventional PT in Diabetic Population)
- Spine Mobilization With Leg Movement+ Conventional PT in non Diabetic Population) (Experimental): The therapist will be applying transverse glide at spinous process towards floor. Other Therapist extended with slight abduction of 10 degrees and hip and knee flexed to 45 degrees. The participant will actively move into SLR with other therapist assistance. If participant feel pain, then ask them to breathe deeply and hold position for 3 sec.
  Interventions: Other: SMWLM+ Conventional PT in non Diabetic Population)

INTERVENTIONS:
Other: CLNDT+ Conventional PT in Diabetic Population): — The participant will be asked to sit on edge of table with hand behind the back with neutral spine. Then patient will be asked to adopted slump forward thoracic and lumbar spine. Then flex the patient neck passively and extend the patient asymptomatic knee with ankle dorsiflexion passively. Adopt this position for 30 sec and 12 rep will be perform for 3 sets and 4 rep per set. Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 10 min 2. Hot pack for 15 min 3. Bridging Exercises (10 rep x 1 Set with 3 sec hold) 4. Ankle pumps (10 rep x 1 Set).
  Arms: Contralateral Leg Neuro Dynamic+ Conventional PT in Diabetic Population):
Other: CLNDT+ Conventional PT in non Diabetic Population): — The participant will be asked to sit on edge of table with hand behind the back with neutral spine. Then patient will be asked to adopted slump forward thoracic and lumbar spine. Then flex the patient neck passively and extend the patient asymptomatic knee with ankle dorsiflexion passively. Adopt this position for 30 sec and 12 rep will be perform for 3 sets and 4 rep per set. Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 10 min 2. Hot pack for 15 min 3. Bridging Exercises (10 rep x 1 Set with 3 sec hold) 4. Ankle pumps (10 rep x 1 Set).
  Arms: contralateral Leg Neuro Dynamic+ Conventional PT in non Diabetic Population):
Other: SMWLM+ Conventional PT in Diabetic Population) — the participant will be asked to adopt side-lying position on their un-effected side, at edge of treatment table. Then The therapist will be applying transverse glide at spinous process towards floor. Other Therapist extended with slight abduction of 10 degrees and hip and knee flexed to 45 degrees. The participant will actively move into SLR with other therapist assistance. If participant feel pain, then ask them to breathe deeply and hold position for 3 sec. Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 10 min 2. Hot pack for 15 min 3. Bridging Exercises (10 rep x 1 Set with 3 sec hold) 4. Ankle pumps (10 rep x 1 Set).
  Arms: Spine Mobilization With Leg Movement+ Conventional PT in Diabetic Population)
Other: SMWLM+ Conventional PT in non Diabetic Population) — the participant will be asked to adopt side-lying position on their un-effected side, at edge of treatment table. Then The therapist will be applying transverse glide at spinous process towards floor. Other Therapist extended with slight abduction of 10 degrees and hip and knee flexed to 45 degrees. The participant will actively move into SLR with other therapist assistance. If participant feel pain, then ask them to breathe deeply and hold position for 3 sec. Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 10 min 2. Hot pack for 15 min 3. Bridging Exercises (10 rep x 1 Set with 3 sec hold) 4. Ankle pumps (10 rep x 1 Set).
  Arms: Spine Mobilization With Leg Movement+ Conventional PT in non Diabetic Population)

SUMMARY:
The aim of this randomized clinical trial is to find the comparison of CLNDT and SMWLM technique in diabetic and non-diabetic sciatica patients on reducing back pain and improving range of motion of knee

DETAILED DESCRIPTION:
Sciatica is the broad term describe as radicular pain/ or paresthesia that originate from low back and radiate along sciatic nerve or with associated lumbosacral nerve root. Sciatica may occur unilaterally or bilaterally with or without lower extremity pain, People with sciatica describe sharp aching and radiating leg pain. It may cause neurological problem such as weakness, numbness or hypo-reflexes and in some cases bladder dysfunction may be present. Pain and discomfort in sciatica affect daily life activities such as walking, bending and running adversely which affect the quality of life.

Diabetes mellitus is a chronic hyperglycemic multisystem disorder which is characterized by either genetic or metabolic dysfunction. It is further classified into two categories type 1 diabetes mellitus (T1DM) which is genetic disorder that prevents the pancreatic beta cells to secrete insulin either due to destruction or reduced number of pancreatic beta cells and type 2 diabetes mellitus (T2DM) is a metabolic disorder in which peripheral insulin receptors of the body become resistant to insulin. The underlying pathophysiology of diabetes and lumbar spine disorders shows a strong association between lumbar degeneration and type 2 diabetes as there is increasing end product of toxic glycation, Expression of MMP-2 related to degradation of extracellular matrix and hyperglycemia induced inflammation of disc, although these changes were observed in animals as in human there is still some lacking about its pathophysiology.

Contralateral leg neuro-dynamic technique was introduced by Shacklock on Maitland concept of slump test that with in slump test position contralateral leg pain is reduced by maintaining this position. This technique is use to reduced pain and increase ROM in sciatica patients. Spinal Mobilization with leg movement was developed by Brain Mulligan, in this technique continuous lateral glides was applied on spinous process and performing actively or passively leg movement this technique is also use for sciatica patients to reduce pain and increase ROM.

The Rational of present study is to determine which technique CLNDT or SMWLM is more effective than other for Pain, ROM, and disability in diabetic and non- diabetic patients with sciatica. It will also determine effect of HbA1C level on pain, ROM and Disability on CLNDT and SMWLM techniques in Diabetic patients with sciatica

ELIGIBILITY:
Inclusion Criteria:

* Patients having sciatica due to degenerative lumbar spine disorder confirm by Straight leg Rise test and Slump test.
* Patients having unilateral radiating leg pain
* Type 2 Diabetic population with past 3 years' history of Diabetes with HbA1c value 5.7% or above

Exclusion Criteria:

* Subject having bilateral leg pain or Cauda equina syndrome
* History of fracture at lumbar spine
* Patient having history of lumbar spine surgery or in symptomatic leg
* Subject having lower extremity vascular disease, Malignancy and pregnant female
* Participant having steroid therapy with in last 6 months.
* Subject having Hip pathologies like hip OA, tendinitis and Bursitis.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Goniometer | three weeks
  It is a tool used to measure the range of motion of joint (0-180). Positioning plays a vital part in goniometry because it helps to place the joints in a zero starting or neutral position. The examiner stabilizes the proximal joint component and then carefully moves the distal component of the joint through its entire available range of motion until reaching the end feel. By using universal goniometer ROM of knee will be assessed, patient will be in supine lying with both legs on the table, fulcrum of goniometer will be aligned with lateral epicondyle while stationary arm is in align with lateral epicondyle and midline of femur. While moving arm is with lateral malleolus and fibula border, while maintaining same position flexion and extension will be performing and measure.
Numeric Pain Rating Scale | three weeks
  The NPRS is an eleven-point pain impression scale: the patient rates pain from 0 (no aggravation) to 10 (most exceedingly terrible possible pain). Numeric Pain Rating Scale (NPRS), which was used to survey respondents' impression of the degree of pain that they felt. NPRS has been utilized in different examinations for low back pain.
Modified Oswestry low back pain Disability Index | three weeks
  The Modified Oswestry Low back pain disability index is widely used standardized questionnaires used by health professional to evaluate patient disability level in patient with low back pain that how patients low back pain affect daily life activities. ODI consists of 10 different questions each score range from 0-5 from minimum to maximum. The score of each section is summed and then divided into total and multiply by 100.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No